CLINICAL TRIAL: NCT05184998
Title: Description of the Clinical Outcomes of Hospitalized Patients With Heart Failure With Different Serum Potassium Levels: Analysis of Data From the China National Heart Failure Registration Study
Brief Title: Description of the Clinical Outcomes of Hospitalized Patients With Heart Failure With Different Serum Potassium Levels
Acronym: SPLENDID
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: D9484R00002
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Hyperkalemia; Hypokalemia; Heart Failure
Keywords: Hyperkalemia, Hypokalemia, Heart Failure, serum potassium,
MeSH Terms: conditions — Hyperkalemia; Hypokalemia; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypokalemia group: defined as sK range (0, 3.5] mmo/L
- Normokalemia group: defined as sK range (3.5, 5.0] mmo/L
- Hyperkalemia group: defined as sK range (5.0, ~) mmo/L

SUMMARY:
China National Heart Failure Registration Study (CN-HF) is a nationwide, hospital-based, multicentre, prospective registry study sponsored by Ministry of Science and Technology of the People's Republic of China. It is aimed to understand the etiology, clinical features and treatments of in-hospital HF patients in China [3].

At present, there are few studies to describe the clinical outcomes of HF patients with different sK levels in China. Utilizing the CN-HF database, this study is aimed to describe the sK levels of hospitalized HF patients and its impact to the clinical outcomes of patients.

DETAILED DESCRIPTION:
Blood potassium disorders are a common phenomenon in patients with HF, which may be related to complications of HF (such as decreased potassium intake, renal insufficiency) and medical treatment of HF (such as diuretics, ACEi/ ARB) [9]. It is showed that abnormal changes in sK can cause myocardial cell membrane potential instability, increase the risk of malignant arrhythmia, and result in a high mortality rate [10].

Current guidelines in China recommend ACEi/ARBs, β receptor blockers, MRAs, and diuretics for treating HF patients . However, β receptor blockers, ACEi/ARB and MRA can also cause hyperkalemia , which often leads to dose reduction or even discontinuation of the medicines, it affects the patients to benefit from these treatment.

At present, there are few studies to describe the clinical outcomes of HF patients with different sK levels in China. Utilizing the CN-HF database, this study is aimed to describe the sK levels of hospitalized HF patients and its impact to the clinical outcomes of patients.

ELIGIBILITY:
Inclusion Criteria:

* HF patients with sK measurements on admission of hospitalization in CN-HF database will be included in this study.

Exclusion Criteria:

* not available for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Totally 6,950 HF patients with sK measurements on admission of hospitalization in CN-HF database will be included.
Sampling Method: Non-Probability Sample
Enrollment: 6950 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
the percentages of patients experiencing a composite of rehospitalization for worsened HF and CV death | 3 year
  the percentages of patients experiencing a composite of rehospitalization for worsened HF and CV death during study period in hypokalemia group, normokalemia group and hyperkalemia group, will be derived using the number of patients who experienced either rehospitalization for worsened HF or CV death during study period divided by the total number of patients in each groups.

SECONDARY OUTCOMES:
The percentages of patients experiencing rehospitalization for worsened HF | 3 years
  The percentages of patients experiencing rehospitalization for worsened HF during study period in hypokalemia group, normokalemia group and hyperkalemia group will be derived using the number of patients who had experienced rehospitalization for worsened HF during the study period divided by the total number of patients in each group.
The percentages of patients experiencing CV death | 3 years
  The percentages of patients experiencing CV death during study period in hypokalemia group, normokalemia group and hyperkalemia group will be derived using the number of patients who had died due to CV disease during the study period divided by the total number of patients in each group.
The percentages of patients experiencing all-cause death | 3 years
  The percentages of patients experiencing all-cause death during study period in hypokalemia group, normokalemia group and hyperkalemia group will be derived using the number of patients who had died during the study period divided by the total number of patients in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Zhou, PhD, Principal Investigator — Fudan University
Locations (1):
- Research Site, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9484R00002&attachmentIdentifier=6ac34580-b8fa-4d6b-b3e0-54148b8a49f0&fileName=D9484R00002_redacted_CSR_Synopsis.pdf&versionIdentifier=